CLINICAL TRIAL: NCT02613936
Title: Transcranial Direct Current Stimulation for the Treatment of Deficits After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNM HRRC #15-124; 1P20GM109089-01A1 (NIH)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury; Post Concussive Symptoms; Depression; Executive Dysfunction
Keywords: traumatic brain injury; post concussive symptoms; depression; executive dysfunction; brain stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome; Depression | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active anodal tDCS + cognitive training (Experimental): In this arm, patients with mmTBI will undergo 10 sessions of active tDCS x 30 minutes combined with simultaneous cognitive training on consecutive weekdays.
  Interventions: Device: Anodal tDCS; Behavioral: Cognitive training
- Placebo anodal tDCS + cognitive training (Sham Comparator): In this arm, patients with mmTBI will undergo 10 sessions of placebo tDCS x 30 minutes combined with simultaneous cognitive training on consecutive weekdays.
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Device: Anodal tDCS — Anodal tDCS lowers neuronal membrane potentials, leading to increased probability of depolarization from incoming stimuli.
  Arms: Active anodal tDCS + cognitive training
Behavioral: Cognitive training — Cognitive training involves solving executive function tasks on a computer.

SUMMARY:
Patients with mild-moderate traumatic brain injury (TBI) sustained between 3 months and 5 years ago with prolonged postconcussive symptoms will be recruited. On Day 1 of the study they will undergo neuropsychological (NP) testing. They will then undergo 10 days of Left dorsolateral prefrontal (DLPFC) anodal transcranial direct current stimulation (TDCS) (active or sham) combined with cognitive training. On day 10 NP testing will be obtained again. On Day 30, NP testing will be repeated a 3rd time. At 6 months and 1 year, quality of life, depression, and post concussive symptoms will be assessed.

DETAILED DESCRIPTION:
Our long-term goal is to develop safe and effective treatments for symptoms of mild to moderate TBI (mmTBI) that restore patients to higher levels of functioning, decrease disability, and promote brain healing. The objective of this application is to investigate the use of transcranial direct current stimulation (tDCS) to treat symptoms of executive dysfunction and depression in patients with mmTBI. Our central hypotheses are (1) tDCS paired with relevant cognitive training facilitates improves executive function on National Institutes of Health (NIH)-approved neuropsychological measures, (2) tDCS reduces depression scores on NIH Common Data Elements for TBI, (3) that these improvements in emotion and cognition will be detectable up to one year after stimulation, and (4) certain clinical variables will reliably predict response to tDCS. These objectives were formulated based on our clinical experience with Dr. Ronald Yeo (project mentor) characterizing symptomatic patients with mmTBI in the post-acute setting and groundbreaking research led by Dr. Vincent Clark (project mentor) that has demonstrated robust increases in attention and learning with tDCS.

Specific Aim 1: tDCS for executive dysfunction in mmTBI Experiments in this aim will test the hypothesis that in patients with mmTBI, left prefrontal anodal tDCS concurrent with cognitive training for ten consecutive weekdays will result in significantly more improvement in executive function compared to sham stimulation. Patients with cognitive complaints 3 months to 2 years after mmTBI will be recruited from local emergency departments and brain injury clinics. Aim 1.1: tDCS will be paired with computer-based cognitive training tasks of response inhibition, set shifting, and working memory, while executive function will be measured with the NIH Examiner battery before, immediately after, and one month after stimulation. Aim 1.2: Persistence of post-traumatic symptom reduction and quality of life improvement will be assessed with Common Data Elements instruments via telephone interview at 6 months and one year. Aim 1.3: Clinical predictors of tDCS response including injury severity, premorbid intelligence, and post-traumatic symptom burden will be determined with linear mixed-models analysis.

Specific Aim 2: tDCS for depressive symptoms in mmTBI Experiments in this aim will test the hypothesis that left prefrontal anodal tDCS in patients with mmTBI will significantly reduce depressive symptoms compared to sham stimulation. Aim 2.1: Patients will be assessed for symptoms of depression via self-report instruments and clinician-administered scales from NIH Common Data Elements before, immediately after, and one month after the stimulation protocol. Aim 2.2: Persistence of antidepressant benefit will be assessed via telephone interview at 6 months and one year. Aim 2.3: clinical predictors of tDCS response such as injury severity, premorbid intelligence, and symptom burden will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-55
2. TBI with + loss of consciousness (LOC) less than 24 hours
3. injured between 3 months and 5 years ago
4. Glasgow Coma Score (GCS) between 9 and 15 upon emergency department (ED) admission
5. less than 1 week of post-traumatic amnesia (PTA)
6. 1 out of 4 cognitive symptoms on the Neurobehavioral Symptom Inventory (NSI)

Exclusion Criteria:

1. history of neurological disease or seizures
2. history of psychosis
3. history of recent substance dependence (past 2 years)
4. any skull defect
5. presence of any implanted electrical device
6. recent medical instability (within 3 weeks)
7. pregnancy
8. appointment of a legal representative.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2020-08 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Shuttleworth, PhD, Principal Investigator — UNM Center for Brain Recovery and Repair
Locations (1):
- UNM Center for Brain Recovery and Repair, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data on task performance may be requested from the researchers after study completion.

REFERENCES:
- See also: For interested volunteers please visit this webpage for contact information to enroll. — http://www.mrn.org/research/volunteer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrollment was concluded at 40 based on termination of funding.
Period: Overall Study
Arm/Group | Active Anodal tDCS + Cognitive Training | Placebo Anodal tDCS + Cognitive Training
Started | 20 | 20
Completed | 17 | 17
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Active Anodal tDCS + Cognitive Training: In this arm, 40 patients with mmTBI will undergo 10 sessions of active tDCS x 30 minutes combined with simultaneous cognitive training on consecutive weekdays.
  Anodal tDCS: Anodal tDCS lowers neuronal membrane potentials, leading to increased probability of depolarization from incoming stimuli.
  Cognitive training: Cognitive training involves solving executive function tasks on a computer.
- Placebo Anodal tDCS + Cognitive Training: In this arm, 40 patients with mmTBI will undergo 10 sessions of placebo tDCS x 30 minutes combined with simultaneous cognitive training on consecutive weekdays.
  Cognitive training: Cognitive training involves solving executive function tasks on a computer.
- Total: Total of all reporting groups
Arm/Group | Active Anodal tDCS + Cognitive Training | Placebo Anodal tDCS + Cognitive Training | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (12.3) | 35.8 (13.6) | 34.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 8 | 10 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Examiner Score
Description: The NIH Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER) assesses executive function in four different domains, creating a composite score from all domains, ranging from -3.0 to 2.0 with higher scores indicating better outcome.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Anodal tDCS + Cognitive Training | Placebo Anodal tDCS + Cognitive Training
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 0.617 (0.677) | 0.907 (0.659)
  End of Treatment | 0.865 (0.677) | 1.155 (0.669)
  1 month Visit | 1.037 (0.677) | 1.26 (0.659)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Active Anodal tDCS + Cognitive Training | Placebo Anodal tDCS + Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 3/17 | 0/17
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Anodal tDCS + Cognitive Training (N=17) | Placebo Anodal tDCS + Cognitive Training (N=17)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — skin sensation, irritation, or rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT02613936/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT02613936/ICF_001.pdf